CLINICAL TRIAL: NCT00650598
Title: A Multicentre, Double-Blind, Double-Dummy, Randomised Study of the Analgesic Efficacy and Safety of Valdecoxib Compared to Diclofenac Sodium in Patients Undergoing Knee Arthroscopy Procedure for Anterior Cruciate Ligament Reconstruction
Brief Title: A Multicentre, Double-Blind, Double-Dummy, Randomised Study of the Analgesic Efficacy and Safety of Valdecoxib Compared to Diclofenac Sodium in Patients Undergoing Knee Arthroscopy for Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3471039
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Pain, Postoperative
Keywords: anterior cruciate ligament, arthroscopy, knee, post-surgical pain
MeSH Terms: conditions — Pain, Postoperative | interventions — valdecoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 40 mg (two 20-mg tablets) loading dose by mouth on Day 1 followed by 20 mg twice daily (BID) on Days 2-6
  Arms: Arm 1
Drug: diclofenac — diclofenac sodium delayed release tablets 75 mg by mouth twice daily (BID) for 6 days
  Arms: Arm 2

SUMMARY:
To demonstrate non-inferiority of valdecoxib 20 mg twice daily (BID) (with an initial loading dose of 40 mg followed by a second dose of 20 mg on the first day only) with diclofenac sodium delayed release 75 mg BID in analgesic efficacy, in subjects undergoing knee arthroscopy procedure for anterior cruciate ligament (ACL) reconstruction, when administered for 6 (±1) days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone an uncomplicated ACL reconstruction procedure and were in satisfactory health were included in the study
* In addition, they needed to have a baseline pain intensity of ≥ 50 mm on the VAS and "moderate to severe" pain on the categorical scale within 8 hours of the completion of the surgical procedure to be included

Exclusion Criteria:

* Patient was scheduled to undergo any other surgical procedure, along with the orthopedic procedure, that was expected to produce a greater degree of surgical trauma than the orthopedic procedure alone
* The patient was undergoing bilateral knee arthroscopy
* The patient used conventional NSAIDs, COX-2 inhibitors, or Tramadol during the 6 hours preceding surgery, during surgery or subsequent to the end of surgery, until randomization
* The patient received oxaprozin or piroxicam within one week prior to randomization
* The patient was required to take muscle relaxants, tricyclic antidepressants, tranquilizers, sedatives, hypnotics and neuroleptics, in the post operative period after the patient was randomized into the study
* The patient had been treated with patient controlled analgesia subsequent to the end of the surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2004-03; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Pain - Visual Analogue Scale | Days 1-6

SECONDARY OUTCOMES:
Physical examination | Screening and Day 6
Global Evaluation of Study Medication | Days 1-6
Consumption of Rescue Medication | Days 1-6
Modified Brief Pain Inventory - short form | Days 2-6
Adverse events | Days 1-6
Vital signs | Screening, Day 1, and Day 6
Effect on Pain Medication Questionnaire and Health Resource Utilization | Days 2-6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Pfizer Investigational Site, Adelaide, South Australia, Australia
- Hong Kong (2):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Shatin, New Territories
- Malaysia (2):
  - Pfizer Investigational Site, Cheras, Kuala Lumpur
  - Pfizer Investigational Site, Kuala Lumpur, Kuala Lumpur
- New Zealand (3):
  - Pfizer Investigational Site, Auckland
  - Pfizer Investigational Site, Christchurch
  - Pfizer Investigational Site, Wellington
- Philippines (3):
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon
  - Pfizer Investigational Site, Quezon City
- Pfizer Investigational Site, Singapore, Singapore
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (3):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Keelung
  - Pfizer Investigational Site, Taipei
- Pfizer Investigational Site, Bangkok, Thailand
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471039&StudyName=A%20Multicentre%2C%20Double-Blind%2C%20Double-Dummy%2C%20Randomised%20Study%20of%20the%20Analgesic%20Efficacy%20and%20Safety%20of%20Valdecoxib%20Compared%20to%20Diclofenac%20